CLINICAL TRIAL: NCT00320138
Title: Acupuncture for the Treatment of Trauma Survivors
Brief Title: Acupuncture for the Treatment of Posttraumatic Stress Among Military Personnel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Federal government (congressional allocation) (Unknown)
Responsible Party: Principal Investigator, Charles Engel, Dir, Deployment Health Clinical Center, WRNMMC; Associate Professor, psychiatry, USUHS, Uniformed Services University of the Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HO0001-051-0002
Record Dates: First submitted 2006-04-27; First posted 2006-05-03 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
Keywords: PTSD; Posttraumatic Stress; Acupuncture; Randomized Controlled Trial; Complementary medicine; Alternative medicine; Chinese medicine; military healthcare
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture (Active Comparator)
  Interventions: Procedure: Acupuncture, using Chinese Medicine methodology
- Wait List (No Intervention): Usual Care

INTERVENTIONS:
Procedure: Acupuncture, using Chinese Medicine methodology — 4 weeks of 2/week treatments (8 total); 4 standardized and 4 individualized treatments
  Arms: Acupuncture

SUMMARY:
The purpose of this study is to determine the effectiveness of acupuncture as a treatment for Posttraumatic Stress Disorder (PTSD) among military personnel.

DETAILED DESCRIPTION:
Untreated Posttraumatic Stress Disorder (PTSD) leads to decreased force readiness and increased health care utilization. Yet, service members with the disorder may be resistant to traditional treatments or find them undesirable because of side-effects, stigma, and long-term commitment. Acupuncture, which has few known side effects, holds promise as an effective treatment option for PTSD. Acupuncture has been shown to improve well-being and has been successfully used to treat stress, anxiety and pain conditions. In order to test the efficacy of acupuncture for treating the symptoms of PTSD-measured by the PTSD Checklist (PCL)-a 12-week, randomized, waitlist-controlled trial will be conducted using a sample of 75 active duty military personnel. Participants will receive an eight-session acupuncture treatment, and will be evaluated throughout the study by way of clinical assessments and an independent assessing acupuncturist.

ELIGIBILITY:
Inclusion Criteria:

* Active duty military personnel
* Criteria met for PTSD based on Clinician-Administered PTSD Scale (CAPS) interview
* A stable medication dosing regimen or therapeutic treatment schedule for at least eight (8) weeks prior to beginning the study.

Exclusion Criteria:

* Acupuncture treatment within the previous 6 months
* Pain greater than or equal to level 8 on the Numeric Rating Scale for Pain
* Significant head injury with loss of consciousness greater than 1 hour
* Uncontrolled diabetes mellitus: fasting blood glucose >180 mg/dl
* Unstable or uncontrolled endocrine disorders, thyroid disease, renal failure, anemia, hemorrhagic diathesis, renovascular disease, Cushing's disease, or hyperaldosteronism
* Unwillingness on the part of participants to complete all study visits and/or the daily Life Chart
* Pregnancy
* Scheduled surgery during the treatment phase of the study
* Medical instability sufficient to warrant inpatient treatment in the medical or intensive care units
* Psychiatric symptoms sufficient to warrant inpatient treatment by the clinical care team
* Psychosis within the past two years
* A traumatic experience, as defined by the DSM-IV criterion A for ASD/PTSD, within the past 30 days

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2006-03; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist (PCL) | baseline, 1 month, 2 months, and 3 months
  The PCL is a widely used measure of PTSD symptom presence and severity among veterans. It is a 17-item measure that assesses the symptoms of PTSD listed in the DSM-IV. Respondents indicate on a 5-point scale (1-5) the degree to which they have been bothered by each symptom in the past month. The PCL-M yields a total severity score ranging from 17 to 85.

SECONDARY OUTCOMES:
Clinician-Administered PTSD Scale | baseline, 3 months
  The CAPS is a 30 item, clinician-administered structured interview that is often referred to as the "gold standard" for diagnosing PTSD. The CAPS measures PTSD and ASD symptoms (based on the DSM-IV symptom criteria) related to up to three traumatic events. Higher scores indicate more intense and more frequent symptoms of PTSD, while lower scores represent the absence of or less intense, less frequent symptoms of PTSD. The CAPS was used in this study as the primary diagnostic tool for PTSD at entry into the study and at the three-month follow-up, and will help validate scores on the PCL.
The Trauma History Questionnaire | baseline, 3 months
  ]. This 24 item self-report questionnaire was designed to assess lifetime history of exposure to 23 potentially traumatic experiences including crime, disaster, and physical and sexual assaults It also contains an open-ended question for specifying other extraordinarily stressful situations or events. The data acquired using this instrument will be used to provide general data about the study sample. Additionally, the THQ will be administered at the three-month follow-up to assess the occurrence of traumatic events during the course of the study.
SF-36-Revised | baseline, 3 months
  The SF-36-Revised measures eight general health-related concepts, which have been shown to load into distinct physical and mental health clusters in factor analytic studies in the general population. The eight scales within the SF-36-Revised are: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional and Mental Health (psychological distress and psychological well-being).
Beck Depression Inventory | baseline, 1 month, 2 months, 3 months
  The BDI-II is a 21-item self-report measure that evaluates symptoms of depression. Each item is scored on a scale from 0 to 3. Total scores on BDI range from 0 to 63, with scores of less than 15 indicating normal to mild depression, scores of 15 to 30 indicating moderate depression, and scores above 30 constituting severe depression.
Numeric Rating Scale for Pain | baseline, 1 month, 2 months, 3 months
  The NRS directs participants to rate pain intensity using three, 11-point, 0 ("no pain") to 10 ("pain as bad as you can imagine") numeric rating scales. Instructions ask participants to "Please rate your pain by indicating the number that best describes your pain on average in the last 24 hours", pain "at its worst", and "pain at its least". The NRS was used in this study to evaluate the effect of acupuncture on comorbid symptoms of pain.
PTSD Life Chart Method (PTSD-LCM) | tracked daily throughout 3-month study period
  The life-chart method is a means of illustrating the relationship of life events and treatment interventions to the longitudinal course of illness. The PTSD-LCM was designed to prospectively track primary symptoms of PTSD as well as comorbid symptoms on a daily basis. The PTSD-LCM incorporates the Ecological Momentary Assessment method in a paper-and-pencil format.
Alcohol Use Disorder Identification Test | baseline, 3 months
  The AUDIT was developed by the World Health Organization to identify hazardous and harmful alcohol use in adults and to serve as a brief (10-item) screening instrument for excessive drinking. It was intended to identify a broad spectrum of problem drinkers and distinguish them from both hospitalized alcoholics and from normal drinkers. The instrument was modified for our purposes to inquire about participants' behavior since returning from deployment. It was used to evaluate the effect of acupuncture on comorbid symptoms of alcohol abuse.
Diagnostic evaluation by blind assessing acupuncturist | baseline, 1 month
  The Assessing Acupuncturist examined the patient using TCM diagnostic criteria before the first treatment, after the first four (standardized) treatments, and again at the conclusion of treatment (after the four individualized treatments). The Assessing Acupuncturist will be blind to the treatment conditions. Identical diagnostic procedures were used for patients in the treatment group and in the wait list control group. Evaluations by the Assessing Acupuncturist were be audio-recorded to ensure that they remain blind to the treatment conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Charles C Engel, MD, MPH, Principal Investigator — USUHS Dept. of Psychiatry/DoD Deployment Health Clinical Center, Walter Reed National Military Medical Center
Locations (1):
- Deployment Health Clinical Center, WRNMMC/USUHS Dept. of Psychiatry, Bethesda, Maryland, United States